CLINICAL TRIAL: NCT03212300
Title: Plasticity in Recovery From Surgery: The Effects of Exercise "Prehabilitation" on Cognitive and Functional Recovery After Shoulder Replacement in Older Adults
Brief Title: TSA Exercise Prehabilitation in Older Adults
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inadequate data analysis
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1620740
Record Dates: First submitted 2017-07-06; First posted 2017-07-11 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Postoperative Delirium and Delayed Functional Recovery
Keywords: aerobic exercise training; delirium
MeSH Terms: conditions — Emergence Delirium; Delirium | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic Exercise Training (AET) (Active Comparator): 20 sessions of AET over a 4 week period just prior to surgery
  Interventions: Behavioral: Aerobic Exercise Training (AET)
- treatment as usual (No Intervention): standard treatment

INTERVENTIONS:
Behavioral: Aerobic Exercise Training (AET) — 20 sessions of AET over a 4 week period just prior to surgery
  Other Names: High Intensity Interval Training (HIIT)
  Arms: Aerobic Exercise Training (AET)

SUMMARY:
This is a randomized study to examine whether aerobic exercise training (AET) before total shoulder replacement (TSR) surgery reduces the incidence of post-operative delirium (POD) and shorten time to recovery in elderly patients. POD is a form of sudden change in mental function that can be experienced after undergoing surgery.

DETAILED DESCRIPTION:
This randomized clinical trial will determine whether aerobic exercise training (AET) before total shoulder replacement (TSR) surgery reduces the incidence of post-operative delirium (POD) and shortens time to recovery in elderly patients. Delayed recovery affects up to 30% of surgical patients and imposes enormous costs on patients, caregivers, and society. Patients over 65 are four times more likely to experience POD, a form of sudden change in mental function that could be experienced after undergoing surgery. POD is associated with impaired daily functioning, longer hospital stay, more frequent institutionalization, and increased mortality.

Prevention of POD is a high clinical priority. Evidence suggests that an exaggerated inflammatory response contributes to POD. Human studies show that AET may exert anti-inflammatory effects. Furthermore, recent animal data show that AET attenuates the inflammatory response to surgery and prevents associated cognitive dysfunction.

The trial will enroll elderly patients undergoing TSR surgery to examine whether a low-cost intervention before surgery can improve clinical outcomes (reduction in POD and decrease recovery time). The effects of a 4-week AET program, specifically a type known as high-intensity interval training (HIIT), on the incidence of POD and time to recovery from fatigue and functional impairment. We will also analyze patients' immune state before and after surgery with modern techniques (high-dimensional mass cytometry). Understanding the immune-modulatory effects of AET will reveal mechanisms that can be targeted by interventions other than or in addition to exercise, which may benefit patients who are physically disabled or require urgent surgery, and help identify non-surgical diseases that may benefit from exercise.

ELIGIBILITY:
Patients scheduled for total shoulder replacement

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-09-28 (Actual); Primary Completion 2020-08-12 (Actual); Study Completion 2020-08-12 (Actual)

PRIMARY OUTCOMES:
Cognitive Function after surgery | up to hospital discharge (approximately 1 day)
  Cognition will be assessed using the Nursing Delirium Screen (NU-DESC) scale to determine if there is any change
Cognitive Function after surgery | up to 12 weeks post-operatively
  Cognition will be assessed using the Family Confusion Assessment Method (FAM-CAM) questionnaire to determine if there is any change

SECONDARY OUTCOMES:
Functional Recovery after surgery | up to 12 weeks post-operatively
  Functional recovery will be assessed with the Surgery Recovery Scale (SRS).The SRS sensitively and reliably captures changes in individual patients, which allows construction of patient-specific recovery trajectories
CyTOF of blood samples | Before exercise (approximately 4 weeks before surgery), after exercise (on the morning of surgery), and 1 hour, 6 hours, and 24 hours post-surgery.
  Blood samples will be collected prior to the intervention, prior to and after surgery for high dimensional mass cytometry

CONTACTS AND LOCATIONS:
Overall Officials: Mervyn Maze, MB, CHB, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No